CLINICAL TRIAL: NCT06905379
Title: Remineralization Efficacy of Moringa Oleifera Varnish Vs MI Varnish in Initial Carious Lesions Over 6 Months Follow Up: a Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Taha Hanafi Mahmoud, Phd candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Moringa Oleifera-based varnish
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: White Spot Lesions [Initial Caries] on Smooth Surface of Tooth; Moringa Oleifera
Keywords: Moringa Oleifera; MI varnish; white spot lesions; remineralization; DIAGNOdent; Nyvad criteria
MeSH Terms: interventions — flocculant protein MO 2.1, Moringa oleifera; Paint

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moringa Oleifera based varnish (Experimental): Moring Oleifera Varnish application Using a disposable bond brush, the varnish will be painted on the diagnosed surfaces, then the patient will be instructed to avoid brushing or flossing and to avoid hard and sticky food or any products that may contain alcohol (oral rinses, beverages, etc.) for the next 4 hours after application.
  Interventions: Other: Moringa Oleifera
- MI varnish (Active Comparator): MI Varnish application
  The varnish will be applied on the clean surfaces according to manufacturer instructions as follows:
  1. The foil cover of the MI Varnish unit dosage bottle will be peeled-off and MI Varnish will be stirred with the disposable brush before application.
  2. The surfaces will be covered with a thin uniform layer using a disposable bond brush to avoid clumping.
  3. The area will be allowed to become wet to ensure the setting of the varnish.
  Interventions: Other: Varnish

INTERVENTIONS:
Other: Moringa Oleifera — Moring Oleifera Varnish application Using a disposable bond brush, the varnish will be painted on the diagnosed surfaces, then the patient will be instructed to avoid brushing or flossing and to avoid hard and sticky food or any products that may contain alcohol (oral rinses, beverages, etc.) for the next 4 hours after application.
  Arms: Moringa Oleifera based varnish
Other: Varnish — MI Varnish application
  The varnish will be applied on the clean surfaces according to manufacturer instructions as follows:
  1. The foil cover of the MI Varnish unit dosage bottle will be peeled-off and MI Varnish will be stirred with the disposable brush before application.
  2. The surfaces will be covered with a thin uniform layer using a disposable bond brush to avoid clumping.
  3. The area will be allowed to become wet to ensure the setting of the varnish.
  Arms: MI varnish

SUMMARY:
This randomized clinical trial aimed to test the remineralization effect of laboratory prepared Moringa Oleifera based varnish compared to MI varnish (CPP-ACP) on incipient carious lesions. The study could include any of the following participants: age: 25-35 years, males or females, presentation with at least one active WSLs on the study teeth at the start of the study, good oral hygiene, co-operative patients approving to participate in the trial, have sufficient cognitive ability to understand consent procedures. The main question it aims to answer is in patients with initial caries lesions will Moringa Oleifera varnish have same remineralization efficacy as MI Varnish after 6 months follow up? MI varnish will be used as a comparator as it has been shown in many studies to be superior to fluoride varnish with NaF alone in arresting early caries lesions. The active ingredient, CPP-ACP can slowly release, localize and stabilize amorphous calcium, phosphate, and fluoride on the enamel surface which aids in deep mineralization of white spot lesions.

DETAILED DESCRIPTION:
The aim of this randomized clinical trial is to evaluate the remineralization efficacy of Moringa Oleifera varnish in comparison to CPP-ACP Varnish on initial carious lesions over 6 months follow up period The null hypothesis is that there will be no difference in the remineralization effect between Moringa Oleifera varnish and CPP-ACP Varnish on incipient carious lesions after 6 months follow up.

* Study design: Randomized clinical trial.
* Double-blinded (participants and outcome assessors).
* Allocation ratio; 1:1
* Framework: Superiority frame.

PICOTS:

P (Population): patients (25-35 years) with active non-cavitated incipient carious lesions on the facial surface (smooth surface lesion).

I (Intervention): Moringa Oleifera-based varnish C (Comparator): CPP-ACP Varnish

O (Primary Outcome):

Outcomes Measuring device Measuring unit Primary Outcome Remineralization effect DIAGNOdent (Shalaan et al., 2023) Ordinal data (scores) Secondary Outcomes Caries lesion activity assessment Nyvad criteria (Nyvad and Baelum , 2018) Ordinal data (scores)

T (Time):

T0= Baseline T1= after 3 months T2= after 6 months S (Study design): Randomized clinical trial, parallel groups, two arms, superiority trial with 1:1 allocation ratio.

Study settings:

This clinical study will be held in the clinic of Conservative dental department-Faculty of Dentistry Cairo University, Egypt.

Inclusion criteria of participants:

* Age: 25-35 years.
* Males or females.
* Presentation with at least one active WSLs on the study teeth at the start of the study.
* Good oral hygiene.
* Co-operative patients approving to participate in the trial.
* Have sufficient cognitive ability to understand consent procedures.

Exclusion criteria of participants:

* Participants with parafunctional habits or bruxism.
* Participants with dry mouth.
* Participants with systemic diseases or disabilities that may affect participation.
* Heavy smoking.
* Pregnancy.
* Lack of compliance.
* Severe or active periodontal disease.
* Cognitive impairment

Inclusion criteria of teeth:

* Active non-cavitated initial carious lesions (ICDAS 1&2)
* DIAGNOdent score between (8-15)
* Vital teeth with no signs or symptoms of irreversible pulpitis.
* No signs of clinical mobility.
* Teeth with healthy periodontium.

Exclusion criteria of teeth:

* DIAGNOdent score less than 8 and more than 15
* Untreated cavitated lesions or extensive restorations on the facial surfaces of the study teeth
* Intrinsic or extremely heavy extrinsic staining
* Periapical pathosis or signs of pulpal pathology.
* Non-vital tooth.
* Signs of pathological wear.
* Endodontically treated tooth.
* Severe periodontal affection or tooth indicated for extraction. Inclusion criteria
* Active non-cavitated initial carious lesions (ICDAS 1&2)
* DIAGNOdent score between (8-15)
* Vital teeth with no signs or symptoms of irreversible pulpitis.
* No signs of clinical mobility.
* Teeth with healthy periodontium. Exclusion criteria
* DIAGNOdent score less than 8 and more than 15
* Untreated cavitated lesions or extensive restorations on the facial surfaces of the study teeth
* Intrinsic or extremely heavy extrinsic staining
* Periapical pathosis or signs of pulpal pathology.
* Non-vital tooth.
* Signs of pathological wear.
* Endodontically treated tooth.
* Severe periodontal affection or tooth indicated for extraction.

Examination and diagnosis:

Examination and selection of patients will be done according to inclusion and exclusion criteria. For every patient, personal data, medical and dental history will be recorded. Clinical examination of labial surfaces with active initial lesions will be done by mouth mirror and explorer with proper direct illumination after gentle dryness for 5 seconds to assess the color, texture and light reflection. To avoid intra-examiner errors, all subjects will be examined by the same examiner. After clinical inspection and DIAGNOdent examination, all patients with ICDAS score 1&2 and with DIAGNOdent score (8-15) will be included in the study.

Informed Consent: Eligible participants will be informed with the procedure and an informed consent will be signed.

b) Moringa Oleifera-based varnish laboratory preparation: The Moringa Oleifera extract and varnish will be prepared in the National Research Centre (Giza, Egypt). Moringa Oleifera leaves will be collected, washed then dried and grinded. Afterwards, the extract of the dried powder will be prepared through extraction with 80% ethyl alcohol. The combined ethanolic extract will then be evaporated till dryness at 45 °C using rotary evaporator under reduced pressure. The obtained mark will be dissolved in water, frozen and lyophilized to obtain lyophilized dry powder then dental varnish will be prepared at a concentration of 200ml/mg. This concentration is recommended by Younis et al.,(2020) as the more the concentration of loaded Moringa Oleifera extract, the more mineral deposition and remineralization enhancement.

After preparing the varnish, it will be stored in single-use form dark bottles to avoid any possible light interactions, then the varnish will be sterilized using steam autoclave Samaha et al.,(2023).

c) Remineralizing materials application:

Teeth preparation:

Teeth with initial carious lesions will be polished with a fluoride-free prophylaxis paste. Moisture control will be done using an air syringe and high-volume suction.

Moring Oleifera Varnish application Using a disposable bond brush, the varnish will be painted on the diagnosed surfaces, then the patient will be instructed to avoid brushing or flossing and to avoid hard and sticky food or any products that may contain alcohol (oral rinses, beverages, etc.) for the next 4 hours after application.

MI Varnish application

The varnish will be applied on the clean surfaces according to manufacturer instructions as follows:

1. The foil cover of the MI Varnish unit dosage bottle will be peeled-off and MI Varnish will be stirred with the disposable brush before application.
2. The surfaces will be covered with a thin uniform layer using a disposable bond brush to avoid clumping.
3. The area will be allowed to become wet to ensure the setting of the varnish.
4. Patients will be instructed to avoid brushing or flossing and to avoid hard and sticky food or any products that may contain alcohol (oral rinses, beverages, etc.) for the next 4 hours after varnish application.

Outcomes:

Primary outcome: Remineralization efficacy The DIAGNOdent will be used to quantify objectively the white spot lesions. For every patient, measurements with the DIAGNOdent will be performed and calibrated on a sound enamel (incisal one third of the central incisor) before actual readings. The teeth will be scanned carefully with the tip held in contact with the tooth surface and tilted around the measuring site so that fluorescence could be collected from all directions. Maximum reading will be recorded Singh et al.,(2016).

DIAGNOdent scores: Shalaan et al.,(2023)

* Score 1: 0-4 (healthy tooth structure)
* Score 2: 5-10 (outer half enamel caries)
* Score 3: 11-20 (inner half enamel caries)
* Score 4: 21+ (dentin caries).

Secondary outcome: Caries lesion activity assessment Nyvad criteria will be used to detect the carious lesion activity. The Nyvad criteria are visual tactile caries classification system which can assess the caries activity and severity. Nyvad criteria includes all stages of caries from clinically sound surfaces to non-cavitated carious lesions and microcavitated lesions in enamel up to frank cavitations in dentine Nyvad and Baelum (2018).

Lesion activity can be detected through surface topography and texture; an active lesion in enamel is rough upon probing with the tip of a ball ended probe, unlike the inactive lesion which appears to be shiny and smooth upon probing. These surface phenomena are the visual representation of the demineralization activity of the dental biofilm. Due to scattering of light, rough active non-cavitated enamel lesions appear dull to the naked eye, unlike the surfaces of inactive lesions which appears glossy due to specular reflection. Nyvad and Baelum (2018).

Patient Recruitment:

Patients will be recruited by H.T from outpatient clinic of conservative dentistry department in Faculty of Dentistry, Cairo University. Eligible patients will then be recruited to fulfill the eligibility criteria according to participant timeline.

Assignment of interventions

Allocation:

Randomization:

N.O will perform simple randomization by generating numbers from 1 to .. , divided into two groups denoting letter A and B. Randomization will be done using random Sequence Generator, Randomness and Integrity Services Ltd (https://www.random.org/).

Allocation concealment mechanism:

The allocation sequence will be kept with the contributor (N.O) in sealed tight envelopes concealed from the primary investigator. The principal investigator (H.T) will know the allocation of the consented participant just before starting the operative procedures.

Implementation Sequence generation and allocation concealment will be implemented by N.O.

Masking/blinding:

The patients and assessors (A.H. and D.K.) will be blinded to the material assignment while the operator will not be due to the difference in remineralization material presentation.

Data collection, management, and analysis

Data collection methods:

1. Baseline data collection: For every patient, medical and dental history will be taken. Examination charts will be filled by H.T.
2. Outcome data collection: DIAGNOdent and carious lesions activity will be evaluated by two assessors (A.H. & D.K.) at baseline, after 3 and 6 months, if both assessors differ in score, they will discuss, if did not agree a third assessor will resolve the conflict.

Data Management:

Data entry will be accomplished by H.T & revised by N.O All data will be restored on computer and will be encrypted using a password. This is done to allow accurate data entry thorough revision and protect data from being inadvertently used. Data will be backed up on another computer to prevent it from being lost.

Statistical analysis:

Data will be analyzed using MedCalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium). Categorical data will be described as frequency and percentage. Intergroup comparisons between categorical variables will be performed using the chi square test, while intragroup comparisons within each intervention will be performed using Cochran's Q test followed by pairwise multiple comparisons. Continuous data will be presented as mean and standard deviation. Intergroup comparison will be done using independent t test, while intragroup comparison will be performed using repeated measures ANOVA followed by Bonferroni corrected pairwise comparisons. A p-value less than or equal to 0.05 will be considered statistically significant and all tests will be two tailed. Statistical power of the study will be set at 80 % with 95 % confidence level.

Data monitoring

Monitoring:

Supervisors A.H will monitor this study. Their role is to monitor any risk of bias from participants, operator or assessors, monitor blinding of the assessors and monitor patient safety and outstanding benefits or harms.

Harms H.T should inform participants about the possible harms, if present. Participants are allowed to contact the operator at moment through telephone. The data will be reported to A.H Audit In this trial auditing will be done by the supervisors A.H and D.K to assure the quality of the research methods, preventive techniques and interventions.

Ethics and dissemination:

Research ethics approval Application forms for carrying out the clinical trial, checklist, and informed consent of Research Ethics Committee (REC) Faculty of Dentistry, Cairo University will be retrieved and filled, then will be delivered for (REC) committee for approval; this is done to prevent any ethical problems during the study or any harm for any of the participants.

Protocol amendments If a new protocol is to be implemented, a protocol amendment will be submitted. This will include a new version of the protocol, and a brief explanation of the differences compared to previous versions. Additionally, any changes to the existing protocol that impact the safety of participants, scope of investigation, or scientific quality of the trial will be communicated through an amendment with a brief explanation of the modifications. Furthermore, if a new author is to be added to facilitate the study, an amendment will be submitted that includes the investigator's credentials and qualifications, aiming to prevent ghost authorship.

Informed consent The principal investigator is tasked with obtaining and signing the informed consents on the day of enrollment. The model of the Research Ethics Committee (REC) of the Faculty of Oral & Dental Medicine, Cairo University, will be utilized throughout this clinical trial.

Confidentiality Name and personal data of the participants will not appear on the protocol form and will be maintained secured for 5 years after the trial. This is done for the protection of participants' privacy and civil rights.

Declaration of interest There is no conflict of interest, no funding or material supply from any parties.

Access to data Access to final data will be allowed to the operator and main supervisor and co supervisors of the study who are not involved in the assessment of the outcome.

Post-trial care Patients will be followed up after varnish application for 3 and 6 months.

Dissemination policy Full protocol will be published online in Clinicaltrials.gov to avoid repetition and keep the integrity of the research work.

Thesis will be discussed and defended in front of a judgment committee. The study will be published to report the results of this clinical trial.

ELIGIBILITY:
Inclusion Criteria of participants:

* Presentation with at least one active WSLs on the study teeth at the start of the study.
* Good oral hygiene.
* Co-operative patients approving to participate in the trial.
* Have sufficient cognitive ability to understand consent procedures Inclusion criteria of teeth.
* Active non-cavitated initial carious lesions (ICDAS 1&2)
* DIAGNOdent score between (8-15)
* Vital teeth with no signs or symptoms of irreversible pulpitis.
* No signs of clinical mobility.
* Teeth with healthy periodontium.

Exclusion Criteria of participants:

* Participants with parafunctional habits or bruxism.
* Participants with dry mouth.
* Participants with systemic diseases or disabilities that may affect participation.
* Heavy smoking.
* Pregnancy.
* Lack of compliance.
* Severe or active periodontal disease.
* Cognitive impairment

Exclusion criteria of teeth:

* DIAGNOdent score less than 8 and more than 15
* Untreated cavitated lesions or extensive restorations on the facial surfaces of the study teeth
* Intrinsic or extremely heavy extrinsic staining
* Periapical pathosis or signs of pulpal pathology.
* Non-vital tooth.
* Signs of pathological wear.
* Endodontically treated tooth.
* Severe periodontal affection or tooth indicated for extraction.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Remineralization efficacy | baseline, 3 months and 6 months
  The DIAGNOdent will be used to quantify objectively the white spot lesions. For every patient, measurements with the DIAGNOdent will be performed and calibrated on a sound enamel (incisal one third of the central incisor) before actual readings. The teeth will be scanned carefully with the tip held in contact with the tooth surface and tilted around the measuring site so that fluorescence could be collected from all directions. Maximum reading will be recorded Singh et al.,(2016).
  DIAGNOdent scores: Shalaan et al.,(2023)
  * Score 1: 0-4 (healthy tooth structure)
  * Score 2: 5-10 (outer half enamel caries)
  * Score 3: 11-20 (inner half enamel caries)
  * Score 4: 21+ (dentin caries).

SECONDARY OUTCOMES:
Caries lesion activity assessment | baseline, 3 months and 6 months
  Nyvad criteria will be used to detect the carious lesion activity. The Nyvad criteria are visual tactile caries classification system which can assess the caries activity and severity. Nyvad criteria includes all stages of caries from clinically sound surfaces to non-cavitated carious lesions and microcavitated lesions in enamel up to frank cavitations in dentine Nyvad and Baelum (2018).
  Lesion activity can be detected through surface topography and texture; an active lesion in enamel is rough upon probing with the tip of a ball ended probe, unlike the inactive lesion which appears to be shiny and smooth upon probing. These surface phenomena are the visual representation of the demineralization activity of the dental biofilm. Due to scattering of light, rough active non-cavitated enamel lesions appear dull to the naked eye, unlike the surfaces of inactive lesions which appears glossy due to specular reflection. Nyvad and Baelum (2018).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Zohair El-Hoshy, professor at Cairo University, Principal Investigator — Cairo University
Locations (1):
- Hend Taha Hanafi Mahmoud, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younis SH, Obeid RF, Ammar MM. Subsurface enamel remineralization by Lyophilized Moringa leaf extract loaded varnish. Heliyon. 2020 Sep 28;6(9):e05054. doi: 10.1016/j.heliyon.2020.e05054. eCollection 2020 Sep. PMID 33015394
- [Background] Singh S, Singh SP, Goyal A, Utreja AK, Jena AK. Effects of various remineralizing agents on the outcome of post-orthodontic white spot lesions (WSLs): a clinical trial. Prog Orthod. 2016 Dec;17(1):25. doi: 10.1186/s40510-016-0138-9. Epub 2016 Aug 2. PMID 27480987
- [Background] Obeid RF, Ammar MM, Younis SH. Dentinomimetics and cementomimetics of Moringa oleifera leaves extract. Sci Rep. 2023 Nov 7;13(1):19243. doi: 10.1038/s41598-023-46656-1. PMID 37935743
- [Background] Nyvad B, Baelum V. Nyvad Criteria for Caries Lesion Activity and Severity Assessment: A Validated Approach for Clinical Management and Research. Caries Res. 2018;52(5):397-405. doi: 10.1159/000480522. Epub 2018 Mar 5. PMID 29506010
- [Background] Malcangi G, Patano A, Morolla R, De Santis M, Piras F, Settanni V, Mancini A, Di Venere D, Inchingolo F, Inchingolo AD, Dipalma G, Inchingolo AM. Analysis of Dental Enamel Remineralization: A Systematic Review of Technique Comparisons. Bioengineering (Basel). 2023 Apr 12;10(4):472. doi: 10.3390/bioengineering10040472. PMID 37106659
- [Background] Jwa SK. Efficacy of Moringa oleifera Leaf Extracts against Cariogenic Biofilm. Prev Nutr Food Sci. 2019 Sep;24(3):308-312. doi: 10.3746/pnf.2019.24.3.308. Epub 2019 Sep 30. PMID 31608256
- [Background] Essam Eliwa M, Mohamed Y, Hossam E. Enamel remineralisation prospect of Moringa Oleifera hydrogel, eggshell hydrogel versus sodium fluoride varnish on artificially demineralised primary teeth: in vitro study. Acta Odontol Scand. 2024 May 6;83:264-272. doi: 10.2340/aos.v83.40623. PMID 38709122
- [Background] Duarte K, Thomas B, Varma SR, Kamath V, Shetty B, Kuduruthullah S, Nambiar M. Antiplaque Efficacy of a Novel Moringa oleifera Dentifrice: A Randomized Clinical Crossover Study. Eur J Dent. 2022 Oct;16(4):768-774. doi: 10.1055/s-0041-1736418. Epub 2022 Jan 11. PMID 35016231
- [Background] Bakry AS, Abbassy MA. Increasing the efficiency of CPP-ACP to remineralize enamel white spot lesions. J Dent. 2018 Sep;76:52-57. doi: 10.1016/j.jdent.2018.06.006. Epub 2018 Jun 19. PMID 29933004